CLINICAL TRIAL: NCT01777191
Title: Pharmacokinetic Evaluations of Ixekizumab Following Subcutaneous Administration Using Prefilled Syringe or Auto-Injector in Patients With Moderate-to-Severe Plaque Psoriasis
Brief Title: Evaluation of Ixekizumab Using Auto-Injector or Prefilled Syringe in Participants With Moderate to Severe Plaque Psoriasis
Acronym: UNCOVER-A
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14728; I1F-MC-RHBL (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-01-24; First posted 2013-01-28 (Estimated); Results first posted 2016-05-26 (Estimated); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — ixekizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 80 mg Ixekizumab Auto-Injector (Experimental): Ixekizumab administered by two 80 milligram (mg) subcutaneous (SC) injections at Week 0, then one 80 mg SC injection every 2 weeks (Q2W) at week 2, 4, 6, 8 and 10. Starting from Week 12, 80 mg Ixekizumab Prefilled Syringe was administered by one 80 mg SC injection every 4 weeks (Q4W).
  Interventions: Drug: Ixekizumab Auto-Injector
- 80 mg Ixekizumab Prefilled Syringe (Experimental): Ixekizumab administered by two 80 mg SC injections at Week 0, then one 80 mg SC injection Q2W at week 2, 4, 6, 8 and 10. Starting from Week 12, 80 mg Ixekizumab Prefilled Syringe was administered by one 80 mg SC injection Q4W.
  Interventions: Drug: Ixekizumab Prefilled Syringe

INTERVENTIONS:
Drug: Ixekizumab Auto-Injector — Administered SC by auto-injector
  Other Names: LY2439821
  Arms: 80 mg Ixekizumab Auto-Injector
Drug: Ixekizumab Prefilled Syringe — Administered SC by prefilled syringe
  Other Names: LY2439821
  Arms: 80 mg Ixekizumab Prefilled Syringe

SUMMARY:
The purpose of this study is to evaluate the serum concentration of ixekizumab after administration using either prefilled syringe or auto-injector in participants with moderate to severe plaque psoriasis. Treatment period is followed by 40 weeks optional safety extension.

ELIGIBILITY:
Inclusion Criteria:

* Present with chronic plaque psoriasis based on a confirmed diagnosis of chronic psoriasis vulgaris for at least 6 months prior to randomization
* At least 10% Body Surface Area (BSA) of Psoriasis at screening and at randomization
* Static Physician Global Assessment (sPGA) score of at least 3 AND Psoriasis Area and Severity Index (PASI) score of at least 12 at screening and at randomization
* Candidate for phototherapy and/or systemic therapy
* Men must agree to use a reliable method of birth control during the study
* Women must agree to use birth control or remain abstinent during the study and for at least 12 weeks after stopping treatment

Exclusion Criteria:

* Pustular, erythrodermic, and/or guttate forms of psoriasis
* History of drug-induced psoriasis
* Clinically significant flare of psoriasis during the 12 weeks prior to randomization
* Concurrent or recent use of any biologic agent
* Received systemic psoriasis therapy [such as psoralen and ultraviolet A (PUVA) light therapy] or phototherapy within the previous 4 weeks; or had topical psoriasis treatment within the previous 2 weeks prior to randomization
* Cannot avoid excessive sun exposure or use of tanning booths for at least 4 weeks prior to randomization and during the study
* Have participated in any study with interleukin-17 (IL-17) antagonists, including Ixekizumab
* Serious disorder or illness other than plaque psoriasis
* Serious infection within the last 3 months
* Breastfeeding or nursing (lactating) women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2013-03; Primary Completion 2014-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (25):
- United States (22):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Anaheim, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bakersfield, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santa Monica, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ocala, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Atlanta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Newnan, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Arlington Heights, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Evansville, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Louisville, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lake Charles, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Methuen, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Omaha, Nebraska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Newington, New Hampshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., East Windsor, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Albuquerque, New Mexico
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greensboro, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Exton, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wyomissing, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salt Lake City, Utah
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seattle, Washington
- Puerto Rico (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Caguas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ponce

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Result] Callis Duffin K, Bagel J, Bukhalo M, Mercado Clement IJ, Choi SL, Zhao F, Gill A, Pangallo B, Shuler C, Mallbris L, Jackson K. Phase 3, open-label, randomized study of the pharmacokinetics, efficacy and safety of ixekizumab following subcutaneous administration using a prefilled syringe or an autoinjector in patients with moderate-to-severe plaque psoriasis (UNCOVER-A). J Eur Acad Dermatol Venereol. 2017 Jan;31(1):107-113. doi: 10.1111/jdv.13768. Epub 2016 Aug 8. PMID 27500949

RESULTS

PARTICIPANT FLOW:
Groups:
- 80 mg Ixekizumab Prefilled Syringe: Ixekizumab administered via prefilled syringe as two 80 milligrams (mg) subcutaneous (SC) injections at Week 0, then one 80 mg SC injection every two weeks (Q2W) at week 2, 4, 6, 8 and 10, and were then followed in the optional safety extension period from week 12 to week 48 using the prefilled syringe 80 mg dose every 4 weeks (Q4W).
- 80 mg Ixekizumab Auto-Injector: Ixekizumab administered via auto-injector as two 80 mg SC injections at Week 0, then one 80 mg SC once injection Q2W at week 2, 4, 6, 8 and 10, and were then followed in the optional safety extension period from week 12 to week 48 using the prefilled syringe 80 mg dose Q4W.
Period: Treatment Period (Per) (Week 0-Week 12)
Arm/Group | 80 mg Ixekizumab Prefilled Syringe | 80 mg Ixekizumab Auto-Injector
Started | 102 | 102
Completed | 96 | 94
Not Completed | 6 | 8
Not completed — Adverse Event | 2 | 1
Not completed — Entry Criteria Not Met | 1 | 1
Not completed — Protocol Violation | 1 | 2
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Lack of Efficacy | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Period: Safety Extension Per (Week 12-Week 48)
Arm/Group | 80 mg Ixekizumab Prefilled Syringe | 80 mg Ixekizumab Auto-Injector
Started | 94 (Participation in the safety extension period was optional.) | 91 (Participation in the safety extension period was optional.)
Completed | 85 | 78
Not Completed | 9 | 13
Not completed — Adverse Event | 3 | 3
Not completed — Death | 0 | 1
Not completed — Withdrawal by Subject | 4 | 4
Not completed — Lack of Efficacy | 1 | 2
Not completed — Lost to Follow-up | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- 80 mg Ixekizumab Prefilled Syringe: Ixekizumab administered via prefilled syringe as two 80 mg SC injections at Week 0, then one 80 mg SC injection Q2W at week 2, 4, 6, 8 and 10, and were then followed in the optional safety extension period from week 12 to week 48 using the prefilled syringe 80 mg dose Q4W.
- Total: Total of all reporting groups
Arm/Group | 80 mg Ixekizumab Prefilled Syringe | 80 mg Ixekizumab Auto-Injector | Total
Number analyzed (Participants) | 102 | 102 | 204
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.3 (14.53) | 46.8 (13.09) | 46.5 (13.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 31 | 62
  Male | 71 | 71 | 142
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 33 | 29 | 62
  Not Hispanic or Latino | 69 | 73 | 142
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 5 | 18
  White | 82 | 95 | 177
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Puerto Rico | 19 | 20 | 39
  United States | 83 | 82 | 165
Baseline in Psoriasis Area and Severity Index (PASI) [Mean (Standard Deviation); unit: units on a scale] — The PASI combines assessments of the extent of body-surface involvement in 4 anatomical regions (head, trunk, arms, and legs) and the severity of desquamation, erythema, and plaque induration/infiltration (thickness) in each region, yielding an overall score of 0 or no Ps to 72 for the most severe disease.
  units on a scale | 21.05 (9.379) | 17.76 (6.141) | 19.40 (8.078)
Baseline in Static Physician Global Assessment (sPGA) Score [Number; unit: participants] — The sPGA is the physician's determination of the participant's Ps lesions overall at a given time point. The sPGA is recommended as an endpoint to use to assess efficacy in the treatment of Ps (EMEA 2004). Overall lesions are categorized by descriptions for induration, erythema, and scaling. For the analysis of responses, the participant's Ps is assessed at a given time point on a 6-point scale in which 0 = cleared, 1 = minimal, 2 = mild, 3 = moderate; 4 = severe, 5 = very severe.
  participants
    sPGA=3 | 55 | 53 | 108
    sPGA=4, 5 | 47 | 49 | 96
Baseline in Subcutaneous Administration Assessment Questionnaire (SQAAQ) [Mean (Standard Deviation); unit: units on a scale] — SQAAQ is a self-administered questionnaire which provides an assessment of ease of use and confidence with using a device to administer a subcutaneous injection of drug. Participants and injection assistants responded to questionnaire items using a 7-point Likert scale (from "Strongly Disagree" to "Strongly Agree"). 1 represents "Strongly Disagree" and 7 represents "Strongly Agree".
  units on a scale
    Easy for me to learn how to use (n=99,101) | 6.4 (1.08) | 6.7 (0.91) | 6.6 (1.01)
    Easy for me to unlock (n=93,101) | 6.4 (0.94) | 6.7 (1.01) | 6.6 (0.98)
    Easy to hold in hand when I inject dose (n=99,101) | 6.3 (1.27) | 6.6 (0.97) | 6.4 (1.14)
    Easy to inject my dose (n=99,101) | 6.2 (1.32) | 6.6 (1.00) | 6.4 (1.18)
    Easy to know that my dose is complete (n=99,101) | 6.4 (1.20) | 6.7 (0.93) | 6.6 (1.07)
    Easy to store device in refrigerator (n=94, 97) | 6.5 (0.88) | 6.6 (1.00) | 6.5 (0.94)
    Easy to remove needle shield/cover (n=99, 100) | 6.6 (0.67) | 6.6 (1.09) | 6.6 (0.91)
    Easy to pick up (n=99, 100) | 6.7 (0.67) | 6.7 (0.94) | 6.7 (0.81)
    Overall, easy to use (n=99,101) | 6.4 (1.10) | 6.6 (0.99) | 6.5 (1.05)
    Device is stable during injection (n=99, 101) | 6.3 (1.18) | 6.6 (1.06) | 6.5 (1.12)
    Confident in ability to use the device (n=99, 101) | 6.4 (1.16) | 6.7 (1.06) | 6.5 (1.12)
    I am confident my dose is complete (n=98,101) | 6.6 (1.09) | 6.7 (0.89) | 6.6 (0.99)

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Maximum Serum Concentration (Cmax) by Drug Delivery Device
Description: Cmax by drug delivery device (prefilled syringe or auto-injector) of Ixekizumab, after the 160 mg starting dose was administered on Day 0.
Time Frame: Day 2, Day 4, Day 7, Day 10 and Day 14 (prior to Ixekizumab administration)
Population: All randomized participants who received at least 1 dose of study drug and had evaluable PK data for Cmax.
Measure: Geometric Mean (90% Confidence Interval); unit: micrograms/milliliter (µg/mL)
Arm/Group | 80 mg Ixekizumab Prefilled Syringe | 80 mg Ixekizumab Auto-Injector
Number analyzed (Participants) | 94 | 98
micrograms/milliliter (µg/mL) | 15.0 [13.9 to 16.1] | 14.8 [13.8 to 15.9]

2. Primary Outcome: PK: Area Under the Concentration Time Curve From Time Zero to Last Measured Concentration Value (AUC 0-[Tlast]) by Drug Delivery Device
Description: AUC 0-tlast by drug delivery device (prefilled syringe or auto-injector) of Ixekizumab, after the 160 mg starting dose was administered on Day 0. AUC 0-tlast is equal to AUC 0-14 days where the last time point was 14 days ± 24 hours.
Time Frame: Day 2, Day 4, Day 7, Day 10 and Day 14 (prior to Ixekizumab administration)
Population: All randomized participants who received at least 1 dose of study drug and had evaluable PK data for AUC.
Measure: Geometric Mean (90% Confidence Interval); unit: micrograms*day/milliliter (µg*day/mL)
Arm/Group | 80 mg Ixekizumab Prefilled Syringe | 80 mg Ixekizumab Auto-Injector
Number analyzed (Participants) | 94 | 98
micrograms*day/milliliter (µg*day/mL) | 157 [147 to 168] | 154 [144 to 165]

3. Secondary Outcome: PK: Cmax of Ixekizumab by Site of Injection (Arm, Thigh or Abdomen)
Description: Cmax by site of injection of Ixekizumab, after the 160 mg starting dose was administered on Day 0.
Time Frame: Day 2, Day 4, Day 7, Day 10 and Day 14 (prior to Ixekizumab administration)
Population: All randomized participants who received at least 1 dose of study drug and had evaluable PK data for Cmax.
Measure: Geometric Mean (90% Confidence Interval); unit: µg/ml
Arm/Group | 80 mg Ixekizumab Prefilled Syringe | 80 mg Ixekizumab Auto-Injector
Number analyzed (Participants) | 92 | 98
µg/ml
  Arm (n=30, 29) | 14.4 [12.4 to 16.8] | 11.5 [10.1 to 13.0]
  Abdomen (n=34, 32) | 12.7 [11.3 to 14.2] | 15.4 [13.5 to 17.5]
  Thigh (n=28, 37) | 18.5 [17.0 to 20.1] | 17.6 [16.0 to 19.4]

4. Secondary Outcome: PK: AUC 0-tlast by Site of Injection (Arm, Thigh or Abdomen)
Description: AUC 0-tlast by site of injection of Ixekizumab, after the 160 mg starting dose was administered on Day 0. AUC 0-tlast is equal to AUC 0-14 days where the last time point was 14 days ± 24 hours.
Time Frame: Day 2, Day 4, Day 7, Day 10 and Day 14 (prior to Ixekizumab administration)
Population: All randomized participants who received at least 1 dose of study drug and had evaluable PK data for AUC.
Measure: Geometric Mean (90% Confidence Interval); unit: µg*day/mL
Arm/Group | 80 mg Ixekizumab Prefilled Syringe | 80 mg Ixekizumab Auto-Injector
Number analyzed (Participants) | 92 | 98
µg*day/mL
  Arm (n=30, 29) | 151 [131 to 173] | 124 [109 to 142]
  Abdomen (n=34, 32) | 135 [122 to 150] | 159 [140 to 180]
  Thigh (n=28, 37) | 190 [176 to 206] | 178 [163 to 194]

5. Secondary Outcome: PK: Cmax by Body Weight
Description: Cmax by body weight of Ixekizumab, after the 160 mg starting dose was administered on Day 0. Body weight is defined by (Low: <80 kilogram (kg), Medium: 80-100 kg, or High: >100 kg).
Time Frame: Day 2, Day 4, Day 7, Day 10 and Day 14 (prior to Ixekizumab administration)
Population: All randomized participants who received at least 1 dose of study drug and had evaluable PK data for Cmax.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Groups:
- 80 mg Ixekizumab: Ixekizumab administered via prefilled syringe and auto-injector as two 80 mg SC injections at Week 0, then one 80 mg SC injection Q2W at week 2, 4, 6, 8 and 10, and were then followed in the optional safety extension period from week 12 to week 48 using the prefilled syringe 80 mg dose Q4W.
Arm/Group | 80 mg Ixekizumab
Number analyzed (Participants) | 192
µg/mL
  Low <80 kg (n=68) | 18.2 [16.9 to 19.5]
  Medium 80-100 kg (n=64) | 15.1 [13.8 to 16.5]
  High >100 kg (n=60) | 11.7 [10.8 to 12.7]

6. Secondary Outcome: PK: AUC 0-tlast by Body Weight
Description: AUC 0-tlast by body weight of Ixekizumab, after the 160 mg starting dose was administered on Day 0. AUC 0-tlast is equal to AUC 0-14 days where the last time point was 14 days ± 24 hours. Body weight is defined by (Low: <80 kg, Medium: 80-100 kg, or High: >100 kg).
Time Frame: Day 2, Day 4, Day 7, Day 10 and Day 14 (prior to Ixekizumab administration)
Population: All randomized participants who received at least 1 dose of study drug and had evaluable PK data for AUC.
Measure: Geometric Mean (90% Confidence Interval); unit: µg*day/mL
Arm/Group | 80 mg Ixekizumab
Number analyzed (Participants) | 192
µg*day/mL
  Low <80 kilograms (kg) (n=68) | 193 [181 to 205]
  Medium 80-100 kg (n=64) | 155 [143 to 168]
  High >100 kg (n=60) | 122 [113 to 132]

7. Secondary Outcome: Percentage of Participants Achieving a ≥75%, ≥ 90% and 100% Improvement in Psoriasis Area and Severity Index (PASI): Efficacy of Ixekizumab in Participants With Moderate to Severe Plaque Psoriasis. Measure: Psoriasis Area and Severity Index (PASI)
Description: PASI combines assessments of the extent of body-surface involvement in 4 anatomical regions (head, trunk, arms, and legs) and the severity of desquamation, erythema, and plaque induration/infiltration (thickness) in each region, yielding an overall score of 0 or no Ps to 72 for the most severe disease. Participants achieving PASI 75, 90, or 100 are defined as having an improvement of at least 75%, 90%, or of 100%, respectively, in the PASI scores compared to baseline.
Time Frame: Week 12
Population: All randomized participants. Participants who did not meet the clinical response criteria or had missing data at Week 12 were considered non-responders for Non-Responder Imputation (NRI) analysis.
Measure: Number; unit: percentage of participants
Arm/Group | 80 mg Ixekizumab Prefilled Syringe | 80 mg Ixekizumab Auto-Injector
Number analyzed (Participants) | 102 | 102
percentage of participants
  PASI 75 | 88.2 | 78.4
  PASI 90 | 76.5 | 62.7
  PASI 100 | 48.0 | 42.2

8. Secondary Outcome: Percentage of Participants With a Static Physician Global Assessment (sPGA) (0,1): Efficacy of Ixekizumab in Participants With Moderate to Severe Plaque Psoriasis. Measure: Static Physician Global Assessment (sPGA)
Description: The sPGA is the physician's determination of the participant's Psoriasis (Ps) lesions overall at a given time point. Lesions were categorized by descriptions for induration, erythema, and scaling. Participant's Ps was assessed as 0 (clear), 1 (minimal), 2 (mild), 3 (moderate), 4 (severe), or 5 (very severe). An sPGA responder was defined as having a post-baseline sPGA score of "0" or "1" with at least a 2-point improvement from baseline.
Time Frame: Week 12
Population: All randomized participants. Participants who did not meet the clinical response criteria or had missing data at Week 12 were considered non-responders for NRI analysis.
Measure: Number; unit: percentage of participants
Arm/Group | 80 mg Ixekizumab Prefilled Syringe | 80 mg Ixekizumab Auto-Injector
Number analyzed (Participants) | 102 | 102
percentage of participants | 80.4 | 73.5

9. Secondary Outcome: Percentage of Participants With a Static Physician Global Assessment (sPGA) (0)
Description: The sPGA is the physician's determination of the participant's Ps lesions overall at a given time point. Lesions were categorized by descriptions for induration, erythema, and scaling. Participant's Ps was assessed as 0 (clear), 1 (minimal), 2 (mild), 3 (moderate), 4 (severe), or 5 (very severe).
Time Frame: Week 12
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | 80 mg Ixekizumab Prefilled Syringe | 80 mg Ixekizumab Auto-Injector
Number analyzed (Participants) | 102 | 102
percentage of participants | 51.0 | 43.1

10. Secondary Outcome: Percentage of Device Operation Failures
Description: Device operation failure (that is, incomplete dose administration) was defined as an event during the treatment period (week 0 to week 12) when the participant indicated that a complete dose of ixekizumab was not delivered and/or the drug delivery device did not perform as expected per the directions for use.
Time Frame: Baseline through Week 12
Population: All randomized participants.
Measure: Number; unit: percentage of incomplete injections
Units Other Than Participants: Injections
Arm/Group | 80 mg Ixekizumab Prefilled Syringe | 80 mg Ixekizumab Auto-Injector
Number analyzed (Participants) | 102 | 102
Number analyzed (Injections) | 680 | 674
percentage of incomplete injections | 0 | 0.3
Statistical Analysis 1: Comparison: 80 mg Ixekizumab Prefilled Syringe vs 80 mg Ixekizumab Auto-Injector; Test type: Superiority or Other; p = 0.248, Fisher Exact

11. Secondary Outcome: Percentage of Participants With Anti-Ixekizumab Antibodies
Description: The percentage of participants with treatment-emergent positive anti-ixekizumab antibodies at anytime post-baseline were summarized by drug delivery device group. Percentage was calculated based on the number of evaluable participants and was calculated by number of participants with treatment-emergent positive anti-ixekizumab antibodies / number of evaluable participants * 100%.
Time Frame: Baseline to Week 12
Population: All randomized participants who received a least 1 dose of study drug during the Treatment Period and had evaluable data.
Measure: Number; unit: percentage of participants
Arm/Group | 80 mg Ixekizumab Prefilled Syringe | 80 mg Ixekizumab Auto-Injector
Number analyzed (Participants) | 102 | 99
percentage of participants | 11.8 | 8.1

12. Secondary Outcome: SQAAQ Item Scores: Quality of Life and Outcome Assessments. Measures: Patient Reported Outcomes (PRO)
Description: The SQAAQ is a self-administered questionnaire which provides an assessment of ease of use and confidence with using a device to administer a subcutaneous injection of drug. Participants and injection assistants responded to questionnaire items using a 7-point Likert scale (from "Strongly Disagree" to "Strongly Agree"). 1 represents "Strongly Disagree" while 7 represents "Strongly Agree". The ease of use and confidence of ixekizumab subcutaneous administrations across drug delivery device groups were evaluated by SQAAQ item scores at each post baseline visit.
Time Frame: Baseline, Week 4 and Week 8
Population: All randomized participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 80 mg Ixekizumab Prefilled Syringe | 80 mg Ixekizumab Auto-Injector
Number analyzed (Participants) | 102 | 102
units on a scale
  Easy for me to learn how to use, Week 4 (n=94, 90) | 6.6 (0.67) | 6.7 (0.86)
  Easy for me to unlock, Week 4 (n=86, 90) | 6.6 (0.81) | 6.8 (0.74)
  Easy to hold in hand, Week 4 (n=94, 90) | 6.6 (0.70) | 6.6 (0.91)
  Easy to inject my dose, Week 4 (n=94, 90) | 6.6 (0.76) | 6.7 (0.83)
  Easy to know dose is complete, Week 4 (n=94, 90) | 6.7 (0.53) | 6.7 (0.79)
  Easy to store in refrigerator, Week 4 (n=91, 88) | 6.7 (0.54) | 6.7 (0.77)
  Easy to remove needle shield, Week 4 (n=94, 90) | 6.6 (0.79) | 6.6 (0.95)
  Easy to pick up, Week 4 (n=94, 90) | 6.8 (0.56) | 6.7 (0.80)
  Overall, easy to use, Week 4 (n=94, 90) | 6.6 (0.70) | 6.7 (0.82)
  Device is stable against skin, Week 4 (n=93, 90) | 6.6 (0.81) | 6.6 (1.05)
  Confident in ability to use, Week 4 (n=94, 90) | 6.7 (0.62) | 6.7 (0.83)
  Confident my dose is complete, Week 4 (n=94, 90) | 6.8 (0.44) | 6.8 (0.71)
  Easy for me to learn how to use, Week 8 (n=89, 92) | 6.7 (0.63) | 6.8 (0.69)
  Easy for me to unlock, Week 8 (n=87, 92) | 6.6 (0.67) | 6.8 (0.69)
  Easy to hold when I inject dose, Week 8 (n=89, 92) | 6.6 (0.67) | 6.7 (0.94)
  Easy to inject my dose, Week 8 (n=89, 92) | 6.5 (0.80) | 6.8 (0.82)
  Easy to know dose is complete, Week 8 (n=89, 92) | 6.7 (0.52) | 6.8 (0.70)
  Easy to store in refrigerator, Week 8 (n=89, 92) | 6.7 (0.62) | 6.8 (0.72)
  Easy to remove needle shield, Week 8 (n=89, 92) | 6.6 (0.75) | 6.7 (0.89)
  Easy to pick up, Week 8 (n=89, 92) | 6.7 (0.63) | 6.8 (0.68)
  Overall, easy to use, Week 8 (n=89, 92) | 6.6 (0.76) | 6.8 (0.74)
  Device is stable against skin, Week 8 (n=88, 92) | 6.6 (0.81) | 6.6 (1.10)
  Confident in ability to use, Week 8 (n=89, 92) | 6.7 (0.77) | 6.8 (0.71)
  Confident my dose is complete, Week 8 (n=89, 92) | 6.7 (0.47) | 6.8 (0.70)

ADVERSE EVENTS:
Groups:
- 80 mg Ixekizumab Prefilled Syringe Treatment Period: Ixekizumab administered via prefilled syringe as two 80 mg SC injections at Week 0, then one 80 mg SC injection Q2W at week 2, 4, 6, 8 and 10, and were then followed in the optional safety extension period from week 12 to week 48 using the prefilled syringe 80 mg dose Q4W.
- 80 mg Ixekizumab Auto-Injector Treatment Period: Ixekizumab administered via auto-injector as two 80 mg SC injections at Week 0, then one 80 mg SC once injection Q2W at week 2, 4, 6, 8 and 10, and were then followed in the optional safety extension period from week 12 to week 48 using the prefilled syringe 80 mg dose Q4W.
- 80 mg Ixe Prefilled Syringe Optional Safety Extension: One 80 mg Ixekizumab administered as an SC injection Q4W.
- Follow Up Period: All participants who received at least 1 dose of Ixekizumab entered the follow-up period.
Arm/Group | 80 mg Ixekizumab Prefilled Syringe Treatment Period | 80 mg Ixekizumab Auto-Injector Treatment Period | 80 mg Ixe Prefilled Syringe Optional Safety Extension | Follow Up Period
Serious Adverse Events (participants affected / at risk) | 3/102 | 4/102 | 9/185 | 1/176
Other Adverse Events (participants affected / at risk) | 12/102 | 10/102 | 24/185 | 0/176
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 80 mg Ixekizumab Prefilled Syringe Treatment Period (N=102) | 80 mg Ixekizumab Auto-Injector Treatment Period (N=102) | 80 mg Ixe Prefilled Syringe Optional Safety Extension (N=185) | Follow Up Period (N=176)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 80 mg Ixekizumab Prefilled Syringe Treatment Period (N=102) | 80 mg Ixekizumab Auto-Injector Treatment Period (N=102) | 80 mg Ixe Prefilled Syringe Optional Safety Extension (N=185) | Follow Up Period (N=176)
Injection site reaction (General disorders) | 8 (12) | 5 (8) | 8 (8) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 5 (5) | 16 (19) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days